CLINICAL TRIAL: NCT00318136
Title: A Pilot Study of Bevacizumab Plus Carboplatin and Paclitaxel in Subjects With Advanced, Previously Untreated, Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Bevacizumab Plus Carboplatin and Paclitaxel in Subjects With Advanced, Previously Untreated, Squamous Non-Small Cell Lung Cancer (BRIDGE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3744g
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Results first posted 2010-04-06 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: BRIDGE; NSCLC; Lung Cancer; Avastin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel

ARMS (1):
- Treated with Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg administered intravenously on Day 1 of each 21- to 28-day cycle, beginning on Cycle 3
Drug: Carboplatin — Dose based on Calvert formula, on Day 1 of each 21- to 28-day cycle for a total of 6 cycles
Drug: Paclitaxel — Dose based on patient's body surface area, on Day 1 of each 21- to 28-day cycle for a total of 6 cycles

SUMMARY:
This is an open-label, single-arm, multicenter pilot study to evaluate the safety and efficacy of carboplatin/paclitaxel+bevacizumab in subjects with locally advanced (Stage IIIb with pleural effusion/pericardial effusion), Stage IV, or recurrent squamous Non-Small Cell Lung Cancer (NSCLC) who have not received prior systemic therapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form(s)
* At least 18 years of age
* Advanced histologically or cytologically confirmed predominant squamous NSCLC
* Subjects with treated brain metastases are eligible if there is no evidence of progression or hemorrhage after treatment of the brain metastasis/metastases
* Prior treatment for CNS disease as deemed appropriate by the treating physician
* ECOG performance status 0, 1, or 2
* Measurable or evaluable disease
* Use of an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study (for women of childbearing potential and sexually active men)

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Adjuvant chemotherapy or prior combined modality therapy (chemotherapy plus radiotherapy) if < 6 months has elapsed from completion of treatment to Day 1, Cycle 1
* Extrathoracic metastases as the only sites of disease
* Active malignancy other than lung cancer
* Current, recent, or planned participation in another experimental drug study
* Untreated brain metastases
* Presence of intrathoracic lesion(s) with any cavitation
* Gross hemoptysis within 3 months prior to Day 1
* In the opinion of the investigator or local radiologist, evidence of tumor that is extending into the lumen of a major blood vessel
* Inadequately controlled hypertension
* Unstable angina or NYHA Grade II or greater CHF
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Myocardial infarction within 6 months prior to Day 1, Cycle 1
* Stroke within 6 months prior to Day 1, Cycle 1
* Active symptomatic peripheral vascular disease within 6 months prior to Day 1, Cycle 1
* History of significant vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Current, ongoing treatment with full-dose warfarin or its equivalent
* Current or recent use of aspirin (>325 mg/day)
* Known hypersensitivity to any components of bevacizumab
* Serious, non-healing wound, ulcer, or bone fracture
* UPC ratio ≥ 1.0
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, Cycle 1, or anticipation of need for major surgical procedure during the course of the study
* Pregnancy or lactation
* Inadequate organ function
* Any other medical conditions (including mental illness or substance abuse) deemed by the clinician to be likely to interfere with a subject's ability to provide informed consent, cooperate, or participate in the study, or to interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Faoro, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated With Bevacizumab: Chemotherapy (carboplatin + paclitaxel) in combination with bevacizumab in intervals of chemotherapy alone (Cycles 1 and 2), chemotherapy + bevacizumab (Cycles 3-6), and bevacizumab alone (Cycles 7 and beyond).
Period: Overall Study
Arm/Group | Treated With Bevacizumab
Started | 47
Completed | 2
Not Completed | 45

BASELINE CHARACTERISTICS:
Arm/Group | Treated With Bevacizumab
Number analyzed (Participants) | 31
Age Continuous [Mean (Standard Deviation); unit: years] — Of the 47 enrolled subjects, 31 met the protocol-specified criteria and received bevacizumab.
  years | 65.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Of the 47 enrolled subjects, 31 met the protocol-specified criteria and received bevacizumab.
  Participants
    Female | 10
    Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade ≥3 Pulmonary Hemorrhage Adverse Events
Description: To estimate the rate of National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE), Version 3.0, Grade ≥3 pulmonary hemorrhage adverse events. Per NCI CTCAE v.3: "Grade 3 = Transfusion, interventional radiology, endoscopic, or operative intervention indicated; radiation therapy (i.e., hemostasis of bleeding site); Grade 4 = Life-threatening consequences; major urgent intervention indicated; Grade 5 = Death."
Time Frame: First bevacizumab administration until 60 days after discontinuation of bevacizumab or death
Population: Safety-evaluable patients
Measure: Number; unit: Percentage of patients
Arm/Group | Treated With Bevacizumab
Number analyzed (Participants) | 31
Percentage of patients | 3.2
Statistical Analysis 1: Comparison: Treated With Bevacizumab; Test type: Superiority or Other; Blyth-Still-Casella; Percentage of patients = 3.2, 90% CI [0.3 to 13.5]

2. Secondary Outcome: Selected Adverse Events
Description: Selected treatment-emergent adverse events for any grade of pulmonary hemorrhage, any grade of non-pulmonary hemorrhage, any grade of gastrointestinal perforation, Grade ≥ 2 arterial thromboembolic events, Grade ≥ 2 left ventricular systolic dysfunction, Grade ≥ 3 proteinuria, and Grade ≥ 3 hypertension. Refer to NCI CTCAE v.3 for grading definitions.
  Serious adverse events (SAEs) occurring in any of the above categories are included. See the Serious Adverse Events section below for full SAE reporting.
Time Frame: First bevacizumab administration until 60 days after discontinuation of bevacizumab or death
Population: Safety-evaluable patients
Measure: Number; unit: Patients
Arm/Group | Treated With Bevacizumab
Number analyzed (Participants) | 31
Patients
  Any grade of pulmonary hemorrhage | 2
  Any grade of non-pulmonary hemorrhage | 0
  Any grade of gastrointestinal perforation | 0
  Grade ≥ 2 arterial thromboembolic events | 2
  Grade ≥ 2 left ventricular systolic dysfunction | 1
  Grade ≥ 3 proteinuria | 1
  Grade ≥ 3 hypertension | 5

3. Secondary Outcome: Adverse Events That Led to Discontinuation of Bevacizumab
Description: Any treatment-emergent adverse event leading to study treatment discontinuation
Time Frame: First bevacizumab administration until 60 days after discontinuation of bevacizumab or death
Population: Safety-evaluable patients
Measure: Number; unit: Patients
Arm/Group | Treated With Bevacizumab
Number analyzed (Participants) | 31
Patients
  Cerebral Infarction | 1
  Cerebral Ischemia | 1
  Neuropathy Peripheral | 1
  Deep Vein Thrombosis | 2
  Hypertension | 1
  Dyspnea | 1
  Pulmonary Embolism | 1
  Cardiac Failure Congestive | 1
  Proteinuria | 1

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from enrollment to the time of documented disease progression or death from any cause, whichever occurred earlier. PFS was determined for only those patients that received bevacizumab.
  Summary of PFS (median) was estimated from Kaplan-Meier curve. The 95% confidence interval (CI) for the median was computed using the method of Brookmeyer and Crowley.
Time Frame: Length of study
Population: Enrolled patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treated With Bevacizumab
Number analyzed (Participants) | 31
Months | 6.2 [5.32 to 7.62]

ADVERSE EVENTS:
Arm/Group | Treated With Bevacizumab
Serious Adverse Events (participants affected / at risk) | 18/31
Other Adverse Events (participants affected / at risk) | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated With Bevacizumab (N=31)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Basal Ganglia Infarction (Nervous system disorders) | 1
Cerebral Infarction (Nervous system disorders) | 1
Cerebral Ischemia (Nervous system disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Atrial Flutter (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Confusional State (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated With Bevacizumab (N=31)
Hypertension (Vascular disorders) | 6
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 2
Sinusitis (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.